CLINICAL TRIAL: NCT06625788
Title: CARACTERIZACIÓN CLÍNICA Y ENDOSCÓPICA DE PACIENTES CON MÚLTIPLES ADENOMAS COLORRECTALES: ESPAPOLIP
Brief Title: Clinical and Endoscopic Characterization of Patients With Multiple Colorectal Adenomas: A Multicenter Study in Spain (ESPAPOLYP Study)
Acronym: ESPAPOLYP
Status: Not yet recruiting | Type: Observational
Sponsor: Asociación Española de Gastroenterología (Other)
Responsible Party: Sponsor
Other Study IDs: ESPAPOLYP; MULTIPLE COLORECTAL ADENOMA SP (Other: SPANISH ASSOCIATION OF GASTROENTEROLOGY)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer Control and Prevention
Keywords: polyp; polyposis; colorectal polyposis; multiple colorectal adenoma; colorectal cancer
MeSH Terms: conditions — Polyps; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with 10 or more colorectal adenomas: patients with 10 or more cumulative colorectal adenomas histologically confirmed

SUMMARY:
The aim is to clinically, endoscopically, and molecularly characterize patients with multiple colorectal adenomas, establish the indication for genetic testing to rule out hereditary syndromes and identify the genes to be included, and improve endoscopic screening recommendations for these patients and their relatives.

DETAILED DESCRIPTION:
HYPOTHESIS

Better characterization of patients with MAC (multiple adenomatous colorectal polyps) could help identify predictive factors of germline pathogenic variants.

Identifying predictive factors of germline pathogenic variants would help optimize and standardize selection criteria for MAC patients to undergo genetic panel testing.

The identification of extra-colonic manifestations in these patients would help implement relevant screening strategies.

Studying the incidence of advanced neoplasia in surveillance colonoscopies in MAC patients would help optimize the intervals for endoscopic surveillance.

Understanding the risk of developing CRC and/or MAC in first-degree relatives of MAC patients without known germline pathogenic variants would allow the establishment of specific colorectal neoplasia screening in this population.

The use of the FIT (fecal immunochemical test) in CRC and/or MAC screening in first-degree relatives (FDR) of MAC patients could be useful by reducing the rate of unnecessary colonoscopies.

OBJECTIVES

The project is subdivided into the following four subprojects:

SUBPROJECT 1: GENPOLYP PROTOCOL

Objectives:

To assess adherence to clinical practice guidelines for requesting genetic testing.

To determine which clinical practice guideline is most used for requesting genetic testing.

To establish the prevalence of germline pathogenic mutations in patients with MAP (multiple adenomatous polyps).

To evaluate predictive factors of germline pathogenic mutations in patients with MAP.

SUBPROJECT 2: RE-SURVPOLYP

Objectives:

Clinical characterization of the cohort. To evaluate the prevalence of CRC and advanced neoplasia in patients with MAC. To evaluate the prevalence of gastroduodenal manifestations. To evaluate the prevalence of non-gastrointestinal manifestations. To determine the need for colorectal surgery in MAC patients. To assess the prevalence of CRC and advanced neoplasia in post-surgical surveillance.

SUBPROJECT 3: PRO-SURVPOLYP

Objectives:

To establish the post-polypectomy surveillance schedule based on the AEG/SEMFYC guidelines.

To assess the incidence of advanced neoplasia and CRC at 3, 5, and 10 years. To evaluate predictive factors of advanced neoplasia in surveillance colonoscopies.

To assess CRC mortality at 5 and 10 years. To assess the incidence of fundic gland polyps, gastric adenomas, duodenal adenomas, and ampullary adenomas at 3, 5, and 10 years.

To assess the incidence of ampullary and duodenal adenocarcinoma at 3, 5, and 10 years.

To evaluate the prevalence of H. pylori. To establish screening indications for gastroduodenal lesions, appropriate surveillance intervals, and the endoscopic technique to be used.

SUBPROJECT 4: FAMPOLYP Subproject 4.1: RE-FAMPOLYP

Objective:

To describe the clinicopathological characteristics of the cohort. To evaluate the prevalence of MAC in first-degree relatives (FDRs) of patients with multiple colorectal adenomas.

To evaluate the prevalence of CRC in FDRs of MAC patients. To evaluate the prevalence of variants of uncertain significance (VUS) coinciding between FDRs of patients with multiple colorectal adenomas for whom a multigene panel was requested.

Subproject 4.2: PRO-FAMPOLYP

Objectives:

To evaluate the incidence of CRC and advanced neoplasia in FDRs of patients with MAC under endoscopic surveillance at 5 years.

To assess the incidence of MAC diagnosis in FDRs of patients with MAC under endoscopic surveillance at 5 years.

To evaluate the diagnostic accuracy of the FIT test for CRC screening in FDRs of MAC patients.

METHODOLOGY AND WORK PLAN

SUBPROJECT 1: GENPOLYP PROTOCOL Design: Prospective, multicenter, observational study.

Methodology:

Patient Selection:

In this protocol, all patients who are detected with ≥10 adenomas in consecutive colonoscopies or a single colonoscopy and/or surgical specimen (if they have undergone colorectal surgery) who have not previously undergone germline genetic testing via a multigene panel will be prospectively included. Patients from families with a previously identified germline pathogenic mutation, those with inflammatory bowel disease (IBD), and those with low performance status (ECOG 3-4) will be excluded. Patients who, due to cognitive decline, cannot make decisions may be included if their legal guardian authorizes their inclusion.

In these patients, a multigene panel test will be requested, which must include the study of at least the following genes: MLH1, MSH2, PMS2, MSH6, EPCAM, APC, MUTYH, BMPR1A, PTEN, STK11, SMAD4, POLD, POLE, NTHL1, RNF43, BRCA1, BRCA2, GREM1.

Variables to collect:

The following variables will be collected:

Demographics: sex, age, race. Clinical: personal history of neoplasia (type and age of diagnosis, as well as treatment received), comorbidities (according to Charlson index), weight, height, body mass index (BMI), abdominal circumference, hypertension, dyslipidemia, diabetes mellitus.

Medication use: non-steroidal anti-inflammatory drugs (NSAIDs), acetylsalicylic acid (ASA), proton pump inhibitors (PPIs), calcium, vitamin D.

Dietary habits (validated PREDIMED questionnaire, Annex II), smoking, alcohol, other drug use.

Family history of neoplasia (1st and 2nd degree): age of diagnosis, type of neoplasia, and degree of kinship. Amsterdam II and Bethesda criteria will also be collected (Annex III).

Colonoscopy-related variables: number of colonoscopies until diagnosis, interval between colonoscopies, number of adenomas and serrated lesions resected in each colonoscopy.

Histological findings: for each colonoscopy, apart from the number of adenomas and/or serrated polyps, advanced adenomas (≥10 mm, high-grade dysplasia, or in situ adenocarcinoma), advanced serrated lesions (hyperplastic polyp ≥10 mm, sessile serrated lesion ≥10 mm and/or with dysplasia, traditional serrated adenoma), and/or CRC will be specified. If CRC is detected, location, TNM staging, and results from the DNA repair protein system (MMR) immunohistochemistry will be recorded.

Clinical practice guidelines: used for genetic testing request (Table 1). Genes included in the multigene panel and detected findings: pathogenic mutations, likely pathogenic mutations, and variants of uncertain significance (VUS) will be described.

Analysis of results:

SPSS and MedCalc programs will be used to analyze the results. A descriptive study will be conducted to report the prevalence of germline pathogenic mutations, as well as adherence to clinical practice guidelines. The cohort will then be divided into two groups: patients with a germline pathogenic or likely pathogenic variant vs. those without these variants. Univariate logistic regression will be applied to assess predictive factors of pathogenic or likely pathogenic mutations, and all variables with P<0.1 will be included in a multivariate logistic regression analysis. A significance level of P<0.05 will be established

ELIGIBILITY:
Inclusion Criteria:

* 10 or more adenomas
* >18 years

Exclusion Criteria:

* Inhereted condictions
* Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with 10 or more colorectal adenoma in whom heredutary consictions have been previously excluded
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
colorectal cancer incidence | 5 years
  incidence of invasive CRC

CONTACTS AND LOCATIONS:
Locations (1):
- Asociacion Española de Gastroenterologua, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No